CLINICAL TRIAL: NCT02107638
Title: Effect of Osteopathic Manipulative Medicine on Motor Function, Balance, and Neuroprotective Serum Markers in Parkinson Disease
Brief Title: Effect of Osteopathic Manipulative Medicine on Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Principal Investigator, Sheldon Yao, Associate Professor, Chair of the Department of OMM, New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHS-975
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Osteopathic Manipulative Medicine; Falls; Balance; Motor function
MeSH Terms: conditions — Parkinson Disease | interventions — Manipulation, Osteopathic; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMM treatment arm (Experimental): Subject will receive osteopathic manipulative treatment protocol for Parkinson's disease (PARK-OMM), twice a week for 6 weeks.
  Interventions: Procedure: OMM treatment arm
- Counseling (Active Comparator): Subjects will receive counseling sessions weekly to match the face to face time with a physician during the OMM treatment arm. No OMM will be performed during this 6 week counseling study period.
  Interventions: Other: Counseling

INTERVENTIONS:
Procedure: OMM treatment arm — OMM is a gentle hand-on manual therapy. The research team created a protocol coined "PARK-OMM" protocol. These techniques aim to help treat myofascial restrictions and improve joint range of motion.
  Other Names: Osteopathic Manipulative Treatment (OMT); Osteopathic Manipulative Medicine (OMM); PARK-OMM
  Arms: OMM treatment arm
Other: Counseling — Patients will be counseled on Parkinson's Disease related issues including prevention of falls, medications, diet, nutrition, exercise, tai-chi, yoga, meditation, and mental health.
  Arms: Counseling

SUMMARY:
Parkinson's disease (PD) is defined as a progressive disorder of the nervous system that affects the patient's mobility, balance and cognition. Tremor, slowed movements, and rigidity are physical symptoms which contribute to postural and gait abnormalities seen in many PD patients. Other symptoms include loss of balance and restricted range of motion, increasing the risk of falling. Osteopathic manipulative medicine (OMM) is a form of manual treatment provided by osteopathic physicians. This form of treatment aims to help decrease muscle spasms and improve joint range of motion and movement. We are proposing a pilot study to investigate the impact of OMM on balance, motor function, and falling in PD patients. We are also going to screen for serum biomarker changes to investigate the potential effects of OMM. Our research team and institution have experience in providing osteopathic care and physical rehabilitation for PD patients. In this study, balance and motor function will be evaluated for each subject throughout the study period. We will also keep track of the number of falls. Balance will be measured using Sensory Organization Test (SOT) and motor function will be measured using Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Both tools are non-invasive and clinically proven methods for measuring balance and motor function.

DETAILED DESCRIPTION:
Annually, 60,000 people within the United States are diagnosed with PD.1 The cardinal features of PD include resting tremor, rigidity, asymmetric onset, and bradykinesia.2 These characteristics appear to affect balance. Balance is a complex system that involves maintaining posture, facilitating movement, and recovering equilibrium to control one's body within its limits of stability. Balance involves the coordination of vestibular, visual, auditory, motor, and high level premotor systems, many of which are compromised in PD.3 Previous research found that 46% of the PD subjects fell within a three month period, and that 21% of subjects had their first fall during the three month period.4 Postural instability is a hallmark sign of PD that compromises balance control and increases the risk of falling.5,6

Many falls in PD occur because of postural instability and their inability to organize sensory information. The SOT identifies abnormalities in postural control, somatosensory, visual, and vestibular sensory systems. It offers a composite score that is a percentage based on normal age controls. We recently presented an abstract at the World Parkinson's Conference in Montreal, Canada that showed individual's with PD (n=20) who were categorized as fallers, scored lower on the SOT than non-fallers with PD.7

The pathogenesis of PD is a progressive neurologic depletion of dopaminergic neurons from the basal ganglia which manifests as common motor or extrapyramidal signs: tremor, bradykinesia, and rigidity. As the severity of PD progresses there is frequently postural instability and further disability. There have been relatively few studies investigating the effect of OMM on PD patients. One previous research study demonstrated that a single session of osteopathic manipulative medicine protocol on 10 PD subjects improved gait compared to age-matched sham-controls, particularly stride length, cadence, and maximum velocities of upper and lower extremities.8 Other studies on non-PD subjects have shown that OMM can improve subject balance. In a pilot study 20 elderly subjects with OMM protocol applied weekly for four weeks showed an improvement in postural instability, as measured by changes in anterior-posterior and medial-lateral sway on force plate observations.9 OMM has also been shown to improve subjects with dizziness. The outcomes were measured using the SMART Balance Master©. It was found that the composite score on the SMART Balance Master© significantly improved immediately after intervention as well as one week later. (P<.001)10

OMM utilized in improving gait in PD patients addressed muscle hypertonicity and joint motion restrictions by using muscle energy and articulatory techniques for the spine and the extremities.8 OMM techniques that were used to address balance focused on removing muscle spasms and restrictions of the spine and cranium. Based on our experience of treating PD patients in our clinical practice and the improvement of symptoms in the forementioned studies we developed a PARK-OMM protocol to utilize in this study. The protocol starts with a CV4 technique, which helps to address cranial restrictions, and can potentially affect patient's autonomic function.11,12 The protocol then proceeds to address each major spinal region and the extremities by decreasing muscle hypertonicity and increasing joint range of motion with direct OMM articulatory and muscle energy techniques. These techniques were selected due to their document efficacy in improving joint mobility in the general population as well as in PD both in clinical practice and documented prior studies.13

Hypothesis: OMM treatments twice a week over a 6-week period on PD subjects using a defined OMM protocol will produce a prolonged improvement in motor function measured by the Movement Disorders Society's Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and balance measured by the NeurCom SMART Balance Master© Sensory Organization Test (SOT) leading to a reduced number of falls. We are also going to screen for serum biomarker changes to investigate the potential effects of OMM. We expect that the OMM cohort will have significantly improved motor function scores, balance, and an associated decrease in falls. This would help to establish the role of OMM in the treatment of PD. Positive findings may also lead to additional studies investigating how OMM impacts the quality of life in PD patients. It could also promote further investigation on the potential mechanisms of OMM amongst the PD population.

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed with Parkinson's Disease
* Over the age of 40

Exclusion Criteria:

* no clinical diagnosis of Parkinson's Disease
* having other diagnosed neurological diseases or disorders
* being completely wheelchair bound or having physical deformities that would prevent completion of the assessment tools

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2023-04 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Number of falls | 10 week period
  A fall log will be kept for subjects enrolled to see if there is a difference between those treated the OMM protocol or those who do not

SECONDARY OUTCOMES:
Balance | 10 weeks
  Balance will be measured via SOT measurements

OTHER OUTCOMES:
Motor function | 10-weeks
  Motor function will be assessed via UPDRS scores
Serum biomarkers | 6 weeks
  Blood draws at week 1, 3, 6 to compare changes in serum biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Yao, DO, Principal Investigator — NYIT College of Osteopathic Medicine
Locations (1):
- New York Institute of Technology - Academic Health Care Center, Old Westbury, New York, United States

REFERENCES:
- [Background] Wells MR, Giantinoto S, D'Agate D, Areman RD, Fazzini EA, Dowling D, Bosak A. Standard osteopathic manipulative treatment acutely improves gait performance in patients with Parkinson's disease. J Am Osteopath Assoc. 1999 Feb;99(2):92-8. doi: 10.7556/jaoa.1999.99.2.92. PMID 10079641
- [Background] Lopez D, King HH, Knebl JA, Kosmopoulos V, Collins D, Patterson RM. Effects of comprehensive osteopathic manipulative treatment on balance in elderly patients: a pilot study. J Am Osteopath Assoc. 2011 Jun;111(6):382-8. doi: 10.7556/jaoa.2011.111.6.382. PMID 21771924
- [Background] Fraix M, Gordon A, Graham V, Hurwitz E, Seffinger MA. Use of the SMART Balance Master to quantify the effects of osteopathic manipulative treatment in patients with dizziness. J Am Osteopath Assoc. 2013 May;113(5):394-403. PMID 23667193
- [Background] DiFrancisco-Donoghue J, Apoznanski T, de Vries K, Jung MK, Mancini J, Yao S. Osteopathic manipulation as a complementary approach to Parkinson's disease: A controlled pilot study. NeuroRehabilitation. 2017;40(1):145-151. doi: 10.3233/NRE-161400. PMID 27814309